CLINICAL TRIAL: NCT02452866
Title: Multi-center, Prospective, Open-Label Study to Evaluate the Safety of A Single Dose of SYM-1219, a Granule Formulation Containing 2 Grams of Secnidazole, for the Treatment of Women and Postmenarchal Adolescent Girls With Bacterial Vaginosis
Brief Title: Open-Label Study to Evaluate Safety of A Single Dose of SYM-1219
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Symbiomix Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYM-1219-350
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2020-12

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — secnidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYM-1219 (Experimental): All pateints recieved single dose SYM-1219 Containing 2 Grams of Secnidazole
  Interventions: Drug: SYM-1219

INTERVENTIONS:
Drug: SYM-1219 — Administered with 4 ounces of unsweetened applesauce, and 8 ounces of water
  Other Names: Secnidazole

SUMMARY:
This is a Phase 3, multi-center, prospective, open-label study to evaluate the safety of SYM-1219 granules containing 2 grams of secnidazole in women and postmenarchal adolescent girls with bacterial vaginosis.

DETAILED DESCRIPTION:
Approximately 325 patients will be enrolled. Patients determined to be eligible for the study will receive SYM-1219 granules containing 2 grams of secnidazole orally as a single dose.

Patients determined to be eligible at the Baseline visit will receive a single dose of SYM-1219 granules containing 2 grams of secnidazole in 4 ounces of unsweetened applesauce to be self-administered on Day 1. Patients will be contacted by telephone once between Days 8 to 10 to inquire about possible adverse events. A final study visit will occur on Day 21 to 30 to assess the patient for safety.

ELIGIBILITY:
Inclusion Criteria:

* Are adult females or postmenarchal adolescent girls ≥ 12 years of age.
* Are in good general health as confirmed by a medical history and physical examination, with no known medical or mental health conditions that, in the Investigator's opinion, may interfere with study participation.
* Have a negative urine pregnancy test result prior to study treatment initiation. In addition, female patients of childbearing potential must be using an acceptable form of birth control as determined by the Investigator
* Agree to abstain from alcohol for 3 days following study treatment.
* Have a clinical diagnosis of bacterial vaginosis
* Agree not to use vaginal douches or similar products for the duration of the study.

Exclusion Criteria:

* Are pregnant, lactating, or planning to become pregnant during the study.
* Are menstruating or have vaginal bleeding at the Baseline visit (Day 1).
* Are menopausal as determined by the Investigator
* Are suspected clinically (or confirmed diagnostically) of having alternative causes of vaginal symptoms including candidiasis, Chlamydia trachomatis, Trichomonas vaginalis, Neisseria gonorrhoeae or Herpes simplex
* Have active genital lesions, including active Herpes simplex lesions, or other vaginal or vulvar conditions which could confound the interpretation of the clinical response, as determined by the Investigator
* Have consumed any alcohol within 12 hours prior to treatment with study medication.
* Have a history of an abnormal Pap smear which required cervical biopsy or cervical cauterization within 3 months of the Baseline visit (Day 1).
* Have any history of cervical carcinoma or other carcinomas of the vagina or vulva.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Jonesboro, Arkansas
  - La Mesa, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Groton, Connecticut
  - Clearwater, Florida
  - Leesburg, Florida
  - Miami, Florida
  - North Miami, Florida
  - Plantation, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Roswell, Georgia
  - Shawnee Mission, Kansas
  - Baltimore, Maryland
  - Fall River, Massachusetts
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Saginaw, Michigan
  - Plainsboro, New Jersey
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Myrtle Beach, South Carolina
  - Jackson, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- SYM-1219: Females 18 & over (not menopausal) with recurring incidences of bacterial vaginosis
Period: Overall Study
Arm/Group | SYM-1219
Started | 325
Completed | 321
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Baseline Nugent score
Groups:
- SYM-1219 2g: Open-Label Study to Evaluate the Safety of A Single Dose of SYM-1219, a Granule Formulation Containing 2 Grams of Secnidazole, for the Treatment of Women and Postmenarchal Adolescent Girls with Bacterial Vaginosis
Arm/Group | SYM-1219 2g
Number analyzed (Participants) | 325
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 323
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 325
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72
  Not Hispanic or Latino | 249
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Participants With Treatment Emergent Adverse Events and Laboratory Abnormalities
Description: Safety evaluations will be based on the incidence, intensity, and type of AEs of subjects with clinical cure at TOC/EOS (clinical cure basd on amsel + normalization of Nugent score)
Time Frame: 30days
Population: Safety evaluations were based on the incidence, intensity, and type of AEs,vital signs, and clinical safety laboratory results.
Measure: Count of Participants; unit: Participants
Groups:
- SYM-1219: SYM-1219 Containing 2 Grams of Secnidazole
Arm/Group | SYM-1219
Number analyzed (Participants) | 325
Participants
  Patients with 1 or more TEAE | 95
  Pateints with Laboratory Abnormality | 2

ADVERSE EVENTS:
Groups:
- SYM-1219 2g: SYM-1219 2g single oral dose
Arm/Group | SYM-1219 2g
All-Cause Mortality (participants affected / at risk) | 0/321
Serious Adverse Events (participants affected / at risk) | 1/321
Other Adverse Events (participants affected / at risk) | 63/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYM-1219 2g (N=321)
foot burn (Injury, poisoning and procedural complications) | 1 (1)
loss of consciousness (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYM-1219 2g (N=321)
headache (Nervous system disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
dysgeusia (Nervous system disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal odor (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pruritis (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 9
Chlamydia (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0)
Gonorrhea (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0)
Urinary tract infection (Infections and infestations) | 10
Vaginal mycosis (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory (Infections and infestations) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0)
Vaginal candidiasis (Infections and infestations) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 18
Bacterial vaginosis (Infections and infestations) | 3
Genital herpes (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No